CLINICAL TRIAL: NCT03074058
Title: Bioequivalence Study of BAY 77-1931 Orally Disintegrating Tablet - Randomized, Open-label, Two-way Crossover Study to Establish the Bioequivalence Between BAY 77-1931 Orally Disintegrating Tablet 500 mg and Fosrenol Chewable Tablet 500 mg Administered in Japanese Healthy Male Adult Subjects
Brief Title: Bioequivalence Study of BAY 77-1931 Orally Disintegrating Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18060
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosrenol ODT (Lanthanum Carbonate, BAY77-1931) (Experimental): Fosrenol BAY 77-1931 orally disintegrating tablet (ODT) 500 mg in Period 1 (day 1-3) and Fosrenol chewable tablet 500mg in Period 2 (day 4-6). The washout interval between period 1 and 2 will be at least 14 days.
  Interventions: Drug: Fosrenol ODT (Lanthanum Carbonate, BAY77-1931)
- Fosrenol chewable Tablet (Lanthanum Carbonate, BAY77-1931) (Active Comparator): Fosrenol BAY77-1931 chewable tablet in Period 1 and Fosrenol BAY 77-1931 ODT 500 mg in Period 2. The washout interval between period 1 and 2 will be at least 14 days.
  Interventions: Drug: Fosrenol chewable Tablet (Lanthanum Carbonate, BAY77-1931)

INTERVENTIONS:
Drug: Fosrenol ODT (Lanthanum Carbonate, BAY77-1931) — Fosrenol orally disintegrating tablet, ODT (Lanthanum Carbonate, BAY77-1931) 500 mg, TID
  Arms: Fosrenol ODT (Lanthanum Carbonate, BAY77-1931)
Drug: Fosrenol chewable Tablet (Lanthanum Carbonate, BAY77-1931) — Fosrenol chewable Tablet (Lanthanum Carbonate, BAY77-1931) 500mg, TID
  Arms: Fosrenol chewable Tablet (Lanthanum Carbonate, BAY77-1931)

SUMMARY:
The primary objective of this study was to establish the bioequivalence of two different tablet formulations containing BAY77-1931. The secondary objectives of this study were to assess the safety and tolerability, as well as to Investigate the plasma lanthanum concentration after BAY 77-1931 ODT 500 mg administration.

ELIGIBILITY:
Inclusion Criteria:

* Japanese healthy male adult volunteers (age, 20-45 years; BMI, 17.6-26.4 kg/m2)

Exclusion Criteria:

* Regular use of medicines including Chinese herbal drugs
* Clinically relevant findings in the physical examination
* Subject who cannot take the study drug appropriately (e.g. weak biting force, insufficient salivary flow)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2015-08-04 (Actual); Study Completion 2015-08-21 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Daily urinary phosphate excretion (mmol) on each day | 6 days
  Each study drug was administered as multiple dose over 4-days under fed conditions with a washout interval of at least 14 days in between. Twenty four hours urine collection were repeated 5 times from morning on Day -2 to that on Day 4.
Bioequivalence: Average of daily urinary phosphate excretion (mmol) over 3-day dosing period | baseline and over 3-days
  During lanthanum carbonate TID treatment period over 3 days in each period (period 1 = day 1-3; period 2 = day 4-6)

SECONDARY OUTCOMES:
Pharmacodynamics: Daily urinary phosphate excretion (mmol) on Day 3 | 1 day
Plasma lanthanum concentrations (ng/mL) | 6 days
  To measure plasma concentration of lanthanum, 6 mL of blood were collected before the breakfast on Day 1, Day 2, Day 3 and Day 4, and at 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours after administration on Day 4.
Pharmacokinetics: Cmax,md of lanthanum in plasma from pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days
Pharmacokinetics: tmax,md of lanthanum in plasma from pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days
Pharmacokinetics: Cmax,md,norm of lanthanum in plasma from pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days
Pharmacokinetics: AUC(0-tlast)md,norm of lanthanum in plasma from pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days
Pharmacokinetics: t1/2,md of lanthanum in plasmafrom pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days
Number of adverse events as a measure of safety and tolarability | From Day 1, the day of the first study drug administration, in period 1 (day 1-3) to follow up, 7-10 days after the last study drug administration in period 2 (day 4 - 6)
Pharmacokinetics: AUC(0-tlast)md of lanthanum in plasma from pre-administration (Day 4) to 48 hours after the last administration (Day 6) | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Fukuoka, Fukuoka, Japan